CLINICAL TRIAL: NCT05976698
Title: Effects of LSD on Perceptual Decision-making in Healthy Subjects
Brief Title: LSD-Perceptual-Choice-Study
Acronym: LUCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); University Psychiatric Clinics Basel (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023-00763, pk23Sterzer
Record Dates: First submitted 2023-07-24; First posted 2023-08-04 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: LSD Reaction
Keywords: neural and behavioral indicators; serotonergic system; perceptual decision-making
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, cross-over study
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Intervention order: 10 μg LSD - 20 μg LSD - Placebo (Experimental): Each subject will participate in 3 x 5 h study sessions separated by at least 7 days.
  Order of drug administration will be 10 μg LSD - 20 μg LSD - Placebo. Vials will contain either 10μg (Active) or 0 μg LSD (Placebo). Thus, participants will be administered two vials on each study visit. 1. visit: active+placebo; 2. visit: active+active, 3. visit: placebo+placebo.
  Interventions: Drug: LSD 10 μg; Drug: LSD 20 μg; Drug: Placebo
- Intervention order: 10 μg LSD - Placebo - 20 μg LSD (Experimental): Each subject will participate in 3 x 5 h study sessions separated by at least 7 days.
  Order of drug administration will be 10 μg LSD - Placebo - 20 μg LSD. Vials will contain either 10μg (Active) or 0 μg LSD (Placebo). Thus, participants will be administered two vials on each study visit. 1. visit: active+placebo; 2. visit: placebo+placebo, 3. visit: active+active.
  Interventions: Drug: LSD 10 μg; Drug: LSD 20 μg; Drug: Placebo
- Intervention order: 20 μg LSD - 10 μg LSD - Placebo (Experimental): Each subject will participate in 3 x 5 h study sessions separated by at least 7 days.
  Order of drug administration will be 20 μg LSD - 10 μg LSD - Placebo. Vials will contain either 10μg (Active) or 0 μg LSD (Placebo). Thus, participants will be administered two vials on each study visit. 1. visit: active+active; 2. visit: active+placebo, 3. visit: placebo+placebo.
  Interventions: Drug: LSD 10 μg; Drug: LSD 20 μg; Drug: Placebo
- Intervention order: 20 μg LSD - placebo - 10 μg LSD (Experimental): Each subject will participate in 3 x 5 h study sessions separated by at least 7 days.
  Order of drug administration will be 20 μg LSD -placebo - 10 μg LSD. Vials will contain either 10μg (Active) or 0 μg LSD (Placebo). Thus, participants will be administered two vials on each study visit. 1. visit: active+active; 2. visit: placebo+placebo, 3. visit: active+placebo.
  Interventions: Drug: LSD 10 μg; Drug: LSD 20 μg; Drug: Placebo
- Intervention order: placebo - 10 μg LSD - 20 μg LSD (Experimental): Each subject will participate in 3 x 5 h study sessions separated by at least 7 days.
  Order of drug administration will be placebo - 10 μg LSD - 20 μg LSD. Vials will contain either 10μg (Active) or 0 μg LSD (Placebo). Thus, participants will be administered two vials on each study visit. 1. visit: placebo+placebo; 2. visit: active+placebo, 3. visit: active+active.
  Interventions: Drug: LSD 10 μg; Drug: LSD 20 μg; Drug: Placebo
- Intervention order: placebo - 20 μg LSD - 10 μg LSD (Experimental): Each subject will participate in 3 x 5 h study sessions separated by at least 7 days.
  Order of drug administration will be placebo - 20 μg LSD - 10 μg LSD. Vials will contain either 10μg (Active) or 0 μg LSD (Placebo). Thus, participants will be administered two vials on each study visit. 1. visit: placebo+placebo; 2. visit: active+active, 3. visit: active+placebo.
  Interventions: Drug: LSD 10 μg; Drug: LSD 20 μg; Drug: Placebo

INTERVENTIONS:
Drug: LSD 10 μg — 0.5 h after the start of each study session the participants will be administered 10 μg LSD per os in the form of vials containing 1ml 20% EtOH (ethanol).
Drug: LSD 20 μg — 0.5 h after the start of each study session the participants will be administered 20 μg LSD per os in the form of vials containing 1ml 20% EtOH.
Drug: Placebo — 0.5 h after the start of each study session the participants will be administered placebo per os in the form of vials containing 1ml 20% EtOH.

SUMMARY:
The aim of the study is to characterize the effects of low doses of LSD (d-lysergic acid diethylamide) on behavioral and neural indicators of feedback and feedforward signaling in perceptual decision-making.

DETAILED DESCRIPTION:
The study team will subject healthy participants to multiple perceptual decision-making tasks after the administration of low doses of LSD (d-lysergic acid diethylamide) as a pharmacological challenge. The investigators want to illuminate the behavioral and neural effects of psychedelics on prior beliefs and evidence processing. Each subject will participate in 3 x 5 h study sessions separated by at least 7 days. Subjects will be under continuous supervision until approximately 4.5h after substance administration. The participants are asked to perform the following cognitive tasks alongside EEG measurement after administration of either LSD or placebo: Changepoint task, history bias task, surround suppression task, auditory steady-state response paradigm, motor localizer task.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to adhere to the study protocol and sign the consent form
* ≥ 18 and ≤ 65 years of age at Screening
* Body mass index 18-29
* Fluent understanding of German
* Normal or corrected-to-normal vision
* Willingness to not operate a traffic vehicle or heavy machinery 24 hours after substance administration
* Willingness to refrain from taking illicit psychoactive substances, including cannabis, for the duration of the study
* Willingness to not consume more than one alcoholic standard drink the night before the study sessions and not consume alcohol for 24 h after each study session
* Willingness to abstain from xanthine-based liquids from the evenings prior to the study sessions and during the sessions
* Willingness to use effective birth-control throughout the study duration
* Adequate task performance in the decision-making tasks during a practice session in the screening visit

Exclusion Criteria:

* Recent (<30 days) or current participation in another clinical trial
* Women that are pregnant, nursing, or planning to become pregnant during the study period
* Current use of contraindicated/psychoactive medications or illicit drugs
* Lifetime use of classical psychedelics more than 20 times, or any time within the previous two months
* Consumption of >5 cigarettes per day or >20 alcoholic standard drinks per week
* Severe chronic or acute medical condition
* Hypertension (>140/90 mmHg) or hypotension (<85mmHg systolic)
* Current or lifetime major mental health disorder
* Personal or family (first-degree) history of a primary psychotic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Change in changepoint task | three times (once on each of the three test days; interval between test days at least 7 days)
  Using the changepoint task, it is examined how explicit expectations about upcoming stimuli are derived from the perceptual history and how they influence the perceptual decision in a volatile environment.
  The study team utilizes an established computerized task and analysis pipeline including a behavioral modeling strategy based on Bayesian inference. The task requires participants to view a train of stimuli consisting of checkerboards presented on a half-circle gradient either more on the right or more on the left side of a fixation cross. Each checkerboard represents information about whether stimuli are currently more likely to appear on the right or left side of the screen. The participants have to indicate by button press, whether they believe the right or the left side is active. Task difficulty is fixed.
Change in history bias task | three times (once on each of the three test days; interval between test days at least 7 days)
  With the history bias task, the study team investigates how implicit expectations about upcoming stimuli are derived from perceptual history and how they bias perceptual discrimination.
  In each trial, two circular gratings will be presented concurrently on the left and right sides of a fixation cross. After complete stimulus presentation, the participants indicate by button press which of the two gratings they believe had the stronger contrast in the trial (left vs. right). Task difficulty will be adjusted individually using an online quest staircase procedure, such that participants will always perform at their 75% accuracy level.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Sterzer, Prof. Dr., Principal Investigator — University Psychiatric Clinics Basel
Locations (1):
- University Psychiatric Clinics Basel, Basel, Switzerland